CLINICAL TRIAL: NCT05229081
Title: Impact of Pharmacist-led Educational Intervention on Pneumococcal Vaccination Rates in Cancer Patients: A Randomized Controlled Study
Brief Title: Impact of Pharmacist-led Educational Intervention on Pneumococcal Vaccination Rates in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nesligul Ozdemir, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Oz2214836
Record Dates: First submitted 2022-01-14; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Pneumonia, Bacterial; Cancer; Pneumococcal Infections
MeSH Terms: conditions — Pneumonia, Bacterial; Neoplasms; Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine education (Other): The intervention arm refers to the arm in which the pharmacist gives vaccination education.
  Interventions: Behavioral: vaccine education
- Standard of Care (No Intervention): The control arm refers to the arm that includes patients who receive routine health care services without vaccination education provided by the pharmacist.

INTERVENTIONS:
Behavioral: vaccine education — The educational content was developed based on research and expert perspectives and included general information about immunization, pneumonia, and pneumococcal vaccines, as well as vaccine myths. This information was first conveyed to the patients verbally, and then booklets with the same material were handed to them. The Pneumococcal Conjugate Vaccine 13 (PCV13) vaccination was recommended based on Infectious Disease Society of America (IDSA), Advisory Committee on Immunization Practices (ACIP), and national adult immunization guidelines.
  Arms: Vaccine education

SUMMARY:
According to the World Health Organization (WHO), immunization; is defined as making a person immune or resistant to an infectious disease by applying a vaccine (1). The primary indicator of an effective immunization is that adequate vaccination rates have been achieved. The risk of cancer and chronic diseases increases with advancing age, which increases the importance of immunization in adults.

Cancer patients, one of the patient groups for whom adult immunization is a priority and crucial, are subjected to immunosuppressive medications, making them vulnerable to infections. In cancer patients, infections are severe, antimicrobial treatments are sometimes insufficient, leading to morbidity and mortality. One of these infections is pneumococcal disease caused by Streptococcus pneumonia, with high morbidity and mortality in cancer patients. Invasive pneumococcal disease is seen 23-48 times more frequently in cancer patients compared to healthy individuals. In many countries worldwide, the 13-valent pneumococcal conjugate vaccine and the 23-valent polysaccharide pneumococcal vaccine, both developed to prevent pneumonia caused by Streptococcus pneumonia, are successfully used in childhood vaccination programs within the framework of WHO's immunization policies. However, in Turkey, like in the rest of the world, the required adult immunization rates have not been achieved yet. Immunization rates among cancer patients, one of the patient groups for whom adult vaccination is required, remain below the targeted levels. Pharmacists, one of the health professionals, have significant contributions to increasing vaccination rates in adults. According to studies, pharmacists can help raise immunization rates by providing education and information. In Turkey, no study has been conducted to assess the impact of vaccination education on cancer patients' attitudes and actions about the pneumococcal vaccine. This study aimed to determine the impact of pharmacist-led pneumonia and pneumococcal vaccine education on cancer patients' vaccination attitudes, knowledge, and vaccination rates.

ELIGIBILITY:
Inclusion Criteria:The study will involve patients who have all of the following features simultaneously.

* patients who visit medical oncology outpatient clinics,
* patients who are over 18 years old,
* patients who have been diagnosed with cancer for less than two years,
* patients who are in remission stage (as determined by a medical oncologist),
* patients who have never had the pneumococcal vaccine.

Exclusion Criteria:

* patients who could not communicate in Turkish,
* patients who were illiterate,
* patients who had visual/auditory/cognitive impairments,
* patients who had previously received a pneumococcal vaccine recommendation,
* patients who did not know their pneumococcal immunization status
* patients who want to leave the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Vaccination attitude | 3 months after education provision
  changes in the patients' Vaccination Attitudes Examination (VAX )Scale scores (This scale consists of 12 items and four subgroups (mistrust of vaccine benefit, worries about unforeseen future effects, concerns about commercial profiteering, and preference for natural immunity) to be responded on a 6-point Likert scale, and the total score ranges between 12-72. The higher scores indicate the anti-vaccination attitudes of the patients.)
Knowledge about pneumonia and the pneumococcal vaccine | 3 months after education provision
  changes in the patients' Vaccination Knowledge Questionnaire (VKQ) (that consists of 13 questions to be answered as 'yes/no/unknown')
Vaccination behavior | 3 months after education provision
  changes in the patients' vaccination rates (The vaccination status of patients with the pneumococcal vaccine will be asked.)

SECONDARY OUTCOMES:
the relationship between demographic characteristics and pneumococcal vaccination behavior | 3 months after education provision
  determining factors affecting pneumococcal vaccination behavior in patients. Parameters (age, gender, educational status, etc.) that differ statistically between vaccinated and unvaccinated patients will be determined, and then logistic regression will be made for these parameters to determine the factors affecting vaccinating behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Aygin Bayraktar-Ekincioglu, Study Chair — Hacettepe University Faculty of Pharmacy Department of Clinical Pharmacy/Ankara/Turkey
Locations (1):
- Hacettepe University Faculty of Medicine Department of Medical Oncology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
study protocol and results
Supporting Information: Study Protocol, CSR
Time Frame: Starting in January 2023

REFERENCES:
- [Background] Wong A, Marrie TJ, Garg S, Kellner JD, Tyrrell GJ; SPAT Group. Increased risk of invasive pneumococcal disease in haematological and solid-organ malignancies. Epidemiol Infect. 2010 Dec;138(12):1804-10. doi: 10.1017/S0950268810000919. Epub 2010 Apr 30. PMID 20429967
- [Background] Chiou WY, Hung SK, Lin HY, Chen LC, Hsu FC, Tsai SJ, Yu BH, Lee MS, Li CY. Effectiveness of 23-valent pneumococcal polysaccharide vaccine on elderly patients with colorectal cancer: A population-based propensity score-matched cohort study. Medicine (Baltimore). 2019 Dec;98(50):e18380. doi: 10.1097/MD.0000000000018380. PMID 31852152
- [Background] Urun Y, Akbulut H, Demirkazik A, Cay Senler F, Utkan G, Onur H, Icli F. Perception about influenza and pneumococcal vaccines and vaccination coverage among patients with malignancies and their family members. J BUON. 2013 Apr-Jun;18(2):511-5. PMID 23818370
- [Background] Klassing HM, Ruisinger JF, Prohaska ES, Melton BL. Evaluation of Pharmacist-Initiated Interventions on Vaccination Rates in Patients with Asthma or COPD. J Community Health. 2018 Apr;43(2):297-303. doi: 10.1007/s10900-017-0421-9. PMID 28852915
- [Background] Otsuka SH, Tayal NH, Porter K, Embi PJ, Beatty SJ. Improving herpes zoster vaccination rates through use of a clinical pharmacist and a personal health record. Am J Med. 2013 Sep;126(9):832.e1-6. doi: 10.1016/j.amjmed.2013.02.018. Epub 2013 Jul 3. PMID 23830534
- See also: Immunization — http://www.who.int/topics/immunization/en/